CLINICAL TRIAL: NCT01520922
Title: A Phase II, Multi-centre Study Investigating the Safety and Efficacy of Ofatumumab and Bendamustine Combination in Patients With Untreated or Relapsed Chronic Lymphocytic Leukaemia (CLL)
Brief Title: Ofatumumab Plus Bendamustine in Frontline and Relapsed Chronic Lymphocytic Leukaemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115991; 2011-005178-43 (EudraCT Number)
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Leukaemia, Lymphocytic, Chronic
Keywords: Relapsed or Refractory Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; CLL; Cancer; Lymphoid leukemia; Lymphoblastic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Recurrence; Neoplasms; Leukemia, Lymphoid; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ofatumumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab plus bendamustine (Experimental): In this single arm, Phase II study, each patient who is willing to participate and is found eligible according to the inclusion and exclusion criteria will enter the treatment phase. Eligible subjects will be allocated to receive the following study treatments depending upon their previous CLL treatment status: Subjects with Untreated CLL: Up to 6 monthly intravenous infusions of Ofatumumab (Cycle 1: 300 mg Day 1 and 1000 mg Day 8; subsequent Cycles: 1000 mg at Day 1 every 28 days) in combination with up to 6 Cycles of intravenous infusions of bendamustine (90 mg/m2, Days 1 and 2; every 28 Days). Subjects with Relapsed CLL: Up to 6 monthly intravenous infusions of Ofatumumab (Cycle 1: 300 mg Day 1 and 1000 mg Day 8; subsequent Cycles: 1000 mg at Day 1 every 28 days) in combination with up to 6 Cycles of intravenous infusions of bendamustine (70 mg/m2, Days 1 and 2; every 28 Days).
  Interventions: Biological: Ofatumumab; Drug: Bendamustine

INTERVENTIONS:
Biological: Ofatumumab — Ofatumumab (ARZERRA™) is an immunoglobulin G1κ (IgG1κ) human monoclonal antibody that specifically recognises a distinct epitope encompassing both large and small extracellular loops on the human CD20 molecule expressed on B cells and binds to this site with high affinity with a dissociation half-life of approximately 3 hours. Ofatumumab induces more efficient complement-dependent cytotoxicity (CDC) mediated cell lysis in vitro, compared to rituximab, especially in low CD20 density cells.
  Other Names: Arzerra
Drug: Bendamustine — Bendamustine is a cytostatic drug which structurally combines a purine-like benzamidazol nucleus and a bifunctional alkylating nitrogen mustard group.
  Other Names: Bendamustine hydrochloride; Levact; Ribomustin; Treanda

SUMMARY:
This is a Phase II, open label, single arm, multi-centre study investigating the safety and efficacy of ofatumumab plus bendamustine in subjects with untreated or relapsed CLL.

Each subject from the screening phase who is willing to participate in the study and is found eligible according to the inclusion and exclusion criteria will enter the treatment phase and will receive a maximum of 6 Cycles of study treatment (ofatumumab plus bendamustine). All subjects will receive 3 Cycles of study treatment (Cycles 1, 2 and 3). Eligibility to receive study treatment for Cycles 4, 5 and 6 will be assessed following the 3rd Cycle. Subjects who have achieved at least stable disease with acceptable toxicity following 3 Cycles of treatment will be eligible to continue to receive study treatments for a maximum of 3 further Cycles. In case of progressive disease, at, or at any time after the start of Cycle 4, subjects must discontinue further study treatment and move into the study's follow-up period.

During the treatment phase, all eligible subjects will be allocated to receive the following study treatments:

1. Subjects with Untreated CLL: Up to 6 monthly intravenous infusions of ofatumumab (Cycle 1: 300 mg Day 1 and 1000 mg Day 8; subsequent Cycles: 1000 mg at Day 1 every 28 Days) in combination with up to 6 Cycles of intravenously infused bendamustine (90 mg/m2, Days 1 and 2, every 28 Days).
2. Subjects with Relapsed CLL: Up to 6 monthly intravenous infusions of ofatumumab (Cycle 1: 300 mg Day 1 and 1000 mg Day 8; subsequent Cycles: 1000 mg at Day 1 every 28 Days) in combination with up to 6 Cycles of intravenously infused bendamustine (70 mg/m2, Days 1 and 2, every 28 Days).

The studies primary endpoint is overall response rate (ORR) as determined by Investigator evaluation. The ORR is the percentage of subjects achieving an objective response (i.e., partial response or better), using the IWCLL updated NCI-WG guidelines. Response assessments are planned at the following time-points: After 3 Cycles of ofatumumab plus bendamustine treatment, after 6 Cycles of ofatumumab plus bendamustine treatment and after the last dose, if not after 6 cycles, of ofatumumab plus bendamustine treatment.

Follow-up assessments will be performed every 3 months following the last study treatment. The follow-up period will last for a maximum of 3 years. Response evaluation assessments to determine subject response or progression will be performed during the follow-up period, according to the IWCLL updated NCI-WG guidelines. Following progression, only survival status and details concerning the subject's next CLL therapy will be recorded.

DETAILED DESCRIPTION:
This is a Phase II, open label, single arm, multi-centre study investigating the safety and efficacy of ofatumumab plus bendamustine in subjects with untreated or relapsed CLL.

The primary objective of this study is to evaluate the investigator assessed overall response rate (ORR), using the International Workshop for Chronic Lymphocytic Leukaemia (IWCLL) updated National Cancer Institute-sponsored Working Group (NCIWG) guidelines, in two populations i.e., subjects with previously untreated CLL and subjects with relapsed CLL administered ofatumumab plus bendamustine.

Secondary objectives are to evaluate the overall response rate with computed tomography scan (CT scan) assessment, complete response rate with and without CT scan assessment, progression free survival, overall survival, duration of response, safety and tolerability, disease, prognostic and biological marker correlation with clinical response in the two populations i.e., subjects with previously untreated CLL and subjects with relapsed CLL administered ofatumumab plus bendamustine.

Exploratory objectives are to investigate the relationship between genetic variants in host DNA and the efficacy, safety and/or tolerability of ofatumumab.

Each subject from the screening phase who is willing to participate in the study and is found eligible according to the inclusion and exclusion criteria will enter the treatment phase and will receive a maximum of 6 Cycles of study treatment (ofatumumab plus bendamustine). All subjects will receive 3 Cycles of study treatment (Cycles 1, 2 and 3). Eligibility to receive study treatment for Cycles 4, 5 and 6 will be assessed following the 3rd Cycle. Subjects who have achieved at least stable disease with acceptable toxicity following 3 Cycles of treatment will be eligible to continue to receive study treatments for a maximum of 3 further Cycles. In case of progressive disease, at, or at any time after the start of Cycle 4, subjects must discontinue further study treatment and move into the study's follow-up period.

During the treatment phase, all eligible subjects will be allocated to receive the following study treatments:

1. Subjects with Untreated CLL: Up to 6 monthly intravenous infusions of ofatumumab (Cycle 1: 300 mg Day 1 and 1000 mg Day 8; subsequent Cycles: 1000 mg at Day 1 every 28 Days) in combination with up to 6 Cycles of intravenously infused bendamustine (90 mg/m2, Days 1 and 2, every 28 Days).
2. Subjects with Relapsed CLL: Up to 6 monthly intravenous infusions of ofatumumab (Cycle 1: 300 mg Day 1 and 1000 mg Day 8; subsequent Cycles: 1000 mg at Day 1 every 28 Days) in combination with up to 6 Cycles of intravenously infused bendamustine (70 mg/m2, Days 1 and 2, every 28 Days).

Prior to each treatment Cycle, subjects must have an absolute neutrophil count > 1.0 x 109/L, a platelet count > 75 x 109/L, and must have recovered to Grade 1 or baseline from all clinically significant non-hematologic toxicities, other than nausea, vomiting or alopecia. If these retreatment criteria are not met, a treatment delay of up to 28 Days is permitted; thereafter, study treatment with bendamustine and ofatumumab must be discontinued. In cases of delays up to 14 Days, bendamustine treatment should be continued at the same dosage, but in case of a delay between 15-28 Days, the dosage of bendamustine must be reduced to 60 mg/m2 for all subsequent treatment Cycles for subjects recruited to the study with previously untreated CLL and 50 mg/m2 for all subsequent treatment Cycles for subjects recruited to the study with relapsed CLL.

Additionally, if within any Cycle, a subject develops a clinically significant Grade 3/4 non-hematologic toxicity, other than nausea, vomiting or alopecia, an absolute neutrophil count < 1.0 x 109/L, or a platelet count < 50% of the pre-treatment value, the bendamustine dose will also be reduced as stated above for all subsequent treatment Cycles.

Blood samples, lymph node examination, spleen and liver measurements, and constitutional symptom evaluations are performed monthly throughout the treatment phase. A bone marrow examination is required to confirm complete response (CR) at least two months after the final study treatment and when a subject fulfils the IWCLL updated NCI-WG requirements for CR. CT-Scans will also be performed, at least two months after the final study treatment, for subjects achieving a CR or partial response (PR) according to the IWCLL updated NCI-WG requirements. Follow-up assessments will be performed every 3 months following the last study treatment. The follow-up period will last for a maximum of 3 years. Response evaluation assessments to determine subject response or progression will be performed during the follow-up period, according to the IWCLL updated NCI-WG guidelines [Hallek, 2008]. Following progression, only survival status and details concerning the subject's next CLL therapy will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CLL defined by a circulating B-lymphocyte count of greater than or equal to 5,000/uL at study entry or at any time in the past and flow cytometry confirmation of immunophenotype with CD5, CD19, CD20, CD23, CD79b, and surface Ig prior to first dose of study treatment.
* Active disease and indication for treatment based on the IWCLL updated NCI-WG guidelines, defined by presence of at least any one of the following conditions: Evidence of progressive marrow failure as manifested by development or worsening of anaemia and/or thrombocytopenia; Massive (i.e. at least 6 cm below the left costal margin) or progressive or symptomatic splenomegaly; Massive nodes (i.e. at least 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy; Progressive lymphocytosis with an increase of more than 50% over a two-month period or a lymphocyte doubling time of less than 6 months.
* A minimum of any one of the following disease-related symptoms must be present: a. Unintentional weight loss greater than or equal to 10% within the previous six months; b. Fevers greater than 100.5°F (38.0°C) for greater than or equal to 2 Weeks without evidence of infection; Or c. Night sweats for more than 1 month without evidence of infection.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Age greater than or equal to 18 years.
* Signed written informed consent from either the subject, or their legally acceptable representative if the subject is incapable of giving their own consent, prior to performing any study-specific tests or procedures.
* Subjects enrolled into the previously untreated subject cohort must also meet all of the following criteria: No prior treatment for CLL (prior corticosteroid immunosuppression treatment for autoimmune hemolytic anaemia and idiopathic thrombocytopenic purpura (ITP) is permitted); Be considered inappropriate for fludarabine-based therapy for reasons that include, but are not limited to, advanced age or presence of co-morbidities.
* Subjects enrolled into the relapsed subject cohort must also meet the following criteria: Relapsed CLL: defined as a subject who has received at least one prior CLL therapy and previously achieved a complete or partial remission/response lasting at least 6 months.

Exclusion Criteria:

* Refractory CLL: defined as treatment failure (failure to achieve a CR or PR) or disease progression within 6 months of the last anti-CLL therapy.
* Previous autologous or allogeneic stem cell transplantation.
* Active autoimmune hemolytic anaemia (AIHA) and idiopathic thrombocytopenic purpura (ITP) requiring corticosteroid therapy greater than 25 mg prednisone (or equivalent) or chemotherapy.
* Known transformation of CLL (e.g. Richter's).
* Known central nervous system involvement by CLL. Screening laboratory values: Platelets less than 100 x 109/L (unless due to CLL involvement of the bone marrow). Neutrophils less than 1.5 x 109/L (unless due to CLL involvement of the bone marrow). Serum creatinine greater than 1.5 times the upper limit of normal (ULN); subjects with a serum creatinine greater than 1.5 x ULN will be eligible if the calculated creatinine clearance [Cockcroft, 1976] is greater than or equal to 30 mL/min. Total bilirubin greater than 1.5 times ULN (unless due to liver involvement by CLL or Gilbert's disease). Transaminases greater than 2.5 times ULN.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, active Hepatitis C, and known Human Immunodeficiency Virus (HIV) disease. All HIV-positive subjects are excluded from this study, regardless of whether they have an Acquired Immunodeficiency Syndrome (AIDS) defining disease and/or are on antiviral therapy.
* Other past or current malignancy (with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix or breast) unless the tumour was successfully treated with curative intent at least 2 years prior to trial entry.*
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to first study treatment, congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities.*
* History of significant cerebrovascular disease or event with significant symptoms or sequelae.*
* Glucocorticoid use, unless given in doses less than or equal to 25mg/Day prednisone (or equivalent) for less than 7 Days for exacerbations other than CLL (e.g. asthma).*
* Positive serology for Hepatitis B (HB) defined as a positive test for Hepatitis B surface antigen (HBsAg). In addition, if negative for HBsAg but Hepatitis B core antibody (HBcAb) positive, a Hepatitis B Virus (HBV) DNA test will be performed and if positive the subject will be excluded.
* Known or suspected hypersensitivity to ofatumumab or bendamustine that in the opinion of the investigator is a contraindication to their participation in the present study.
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 Weeks prior to first study treatment dose, whichever is longer, or participation in any other interventional clinical study.
* Known or suspected inability to comply with the study protocol.
* Lactating women, women with a positive pregnancy test at Visit 1 or women (of childbearing potential) as well as men with partners of childbearing potential, who are not willing to use adequate contraception from study start through one year following last ofatumumab dose. Adequate contraception is defined as abstinence, oral hormonal birth control, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device, and male partner sterilisation if male partner is sole partner for that subject. For females in the USA, the use of a double barrier method is also considered adequate (condom or occlusive cap plus spermicidal agent).

  * Subjects can participate in the study if in the opinion of the investigator it is thought not to affect the subject's safety, the conduct of the study or the interpretation of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (6):
  - Novartis Investigative Site, Tuscon, Arizona
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Ogden, Utah
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Czechia (4):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Italy (5):
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Novara, Piedmont
  - Novartis Investigative Site, Turin, Piedmont
- Poland (3):
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Wroclaw
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
- Spain (3):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Majadahonda (Madrid)

REFERENCES:
- [Derived] Flinn IW, Panayiotidis P, Afanasyev B, Janssens A, Grosicki S, Homenda W, Smolej L, Kuliczkowski K, Doubek M, Domnikova N, West SL, Chang CN, Barker AM, Gupta IV, Wright OJ, Offner F. A phase 2, multicenter study investigating ofatumumab and bendamustine combination in patients with untreated or relapsed CLL. Am J Hematol. 2016 Sep;91(9):900-6. doi: 10.1002/ajh.24430. Epub 2016 Jul 3. PMID 27222473

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria at Screening were then allocated to one of the following populations: par. with previously untreated CLL or par. with relapsed CLL. A total of 99 par. were enrolled and 97 par. entered the treatment period. Study results do not include the 2 par. that were not treated in this study
Groups:
- Ofatumumab + Bendamustine 90 mg/m^2: Participants with previously untreated CLL received IV infusions of ofatumumab in combination with bendamustine IV infusions for 6 cycles; each cycle comprised of 28 days. Participants received ofatumumab administered at 300 mg on Day 1, 1000 mg on Day 8 of cycle 1 and 1000 mg on Day 1 of cycles 2, 3, 4, 5 and 6. Bendamustine was administered at 90 mg/m^2 on Days 1 and 2 of each cycle (6 cycles).
- Ofatumumab + Bendamustine 70 mg/m^2: Participants with relapsed CLL received IV infusions of ofatumumab in combination with bendamustine IV infusions for 6 cycles; each cycle comprised of 28 days. Participants received ofatumumab administered at 300 mg on Day 1, 1000 mg on Day 8 of cycle 1 and 1000 mg on Day 1 of cycles 2, 3, 4, 5 and 6. Bendamustine was administered at 70 mg/m^2 on Days 1 and 2 of each cycle (6 cycles).
Period: Treatment Phase
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Started | 44 | 53
Completed | 39 (Completed 6 Cycles of Study Treatment) | 45 (Completed 6 Cycles of Study Treatment)
Not Completed | 5 | 8
Not completed — Physician Decision | 2 | 1
Not completed — Progression | 0 | 2
Not completed — Adverse Event | 3 | 5
Period: Follow up
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Started | 44 | 45
Completed | 44 | 44
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Survival Follow-up
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Started | 21 | 40
Completed | 20 | 40
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2 | Total
Number analyzed (Participants) | 44 | 53 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (10.11) | 66.5 (9.28) | 65.0 (9.76)
Gender [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 29 | 36 | 65
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 42 | 53 | 95
  White - Arabic/North African Heritage | 1 | 0 | 1
  African American/African Heritage | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response (OR), as Assessed by the Investigator
Description: OR is defined as the number of participants achieving an objective response (complete response [CR], CR with incomplete bone marrow recovery [CRi], partial response [PR], and nodular PR [nPR]), after 3 cycles, after 6 cycles, and after the last dose of ofatumumab and bendamustine treatment. CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly)/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL, LC <4000/µL. nPR: persistent nodules BM.
Time Frame: From the start of study treatment until 3 months after the last dose of study treatment
Population: As-treated subjects (ATS) Population: all participants who received at least one dose of both study drugs (ofatumumab and bendamustine). OR was measured using the International Workshop for CLL (IWCLL) updated National Cancer Institute-sponsored Working Group (NCI-WG) guidelines 2008. The 95% exact binomial confidence interval is for CR+CRi+nPR+PR.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  CR | 19 | 6
  CRi | 2 | 2
  nPR | 4 | 8
  PR | 17 | 23
Statistical Analysis 1: Comparison: Ofatumumab + Bendamustine 90 mg/m^2; Test type: Superiority or Other; Percentage of participants = 95, 95% CI 2-sided [84.53 to 99.44] — The estimated value represents the percentage of participants with OR (CR+CRi+nPR+PR) while receiving ofatumumab + bendamustine 90 mg/m^2
Statistical Analysis 2: Comparison: Ofatumumab + Bendamustine 70 mg/m^2; Test type: Superiority or Other; Percentage of participants = 74, 95% CI 2-sided [59.67 to 84.74] — The estimated value represents the percentage of participants with OR (CR+CRi+nPR+PR) while receiving ofatumumab + bendamustine 70 mg/m^2

2. Secondary Outcome: Number of Participants With Overall Response (OR) With Computed Tomography (CT) Scan (CT Scan) Assessment, as Assessed by the Investigator
Description: as for outcome 1
Time Frame: From the start of study treatment until 3 months after the last dose of study treatment
Population: ATS Population. OR was measured using the International Workshop for CLL (IWCLL) updated National Cancer Institute-sponsored Working Group (NCI-WG) guidelines 2008.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  CR | 12 | 5
  CRi | 1 | 2
  nPR | 2 | 6
  PR | 22 | 24

3. Secondary Outcome: Number of Participants With Complete Response (CR) With and Without a CT Scan Assessment After the Last Dose of Study Treatment, as Assessed by the Investigator
Description: Response was determined according to the IWCLL updated NCI-WG guidelines 2008. CR requires all of the following criteria at least 2 months after the last treatment: no lymphadenopathy (Ly)/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500/µL, platelets (PL) >100,000/µL, hemoglobin (Hb) >11.0 g/dL, lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule.
Time Frame: From the start of study treatment until 3 months after the last dose of study treatment
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  CR without CT scan assessment | 19 | 6
  CR with CT scan assessment | 12 | 5

4. Secondary Outcome: Investigator-assessed Kaplan-meier Estimates of Time to Response
Description: Time to response is defined as time from date of the first administration of study treatment to the first response (CR, CRi, nPR, or PR). Response was determined according to the IWCLL updated NCI-WG guidelines 2008. CR: all of the following criteria at least 2 months after last treatment: no lymphadenopathy (Ly)/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11.0 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/ thrombocytopenia/ neutropenia unrelated to CLL but related to drug toxicity. nPR: persistent nodules BM. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11.0 g/dL or 50% improvement over BL, LC <4000/µL.
Time Frame: From the start of study treatment to the first response (CR, CRi, nPR, or PR) (up to 3 Month Follow-up (F/U) visit)
Population: ATS Population. Only participants who had a response (CR, CRi, nPR, or PR) were evaluated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 43 | 47
Months | 0.95 [0.95 to 1.02] | 1.08 [0.95 to 1.87]

5. Secondary Outcome: Investigator-assessed Kaplan-meier Estimates of Duration of Response
Description: The duration of response is defined as the time from the initial response (CR, CRi, nPR, or PR) to the first documented sign of disease progression (PD) or death due to any cause. PD requires at least one of the following: new lesion or increase by >=50% from Baseline in lymphocytes (LC) with at least 5000B-lymphocytes per microliter (5.0 x 10^9/L), lymphadenopathy (Ly), size of liver and spleen, platelets (PL) >= 50% decrease from Baseline, or to <100,000/uL secondary to CLL, hemoglobin (Hb) decrease of >2 g/dL from Baseline or to <10 g/dL secondary to CLL, CLL- transformation, cytopenia after treatment. Response was determined according to the IWCLL updated NCI-WG guidelines 2008.
Time Frame: From time of initial response (CR, CRi, nPR, or PR) to disease progression or death, whichever came first (up to 3 years after the last doseof study treatment)
Population: ATS Population. Only participants with an initial response (CR, CRi, nPR, or PR) with PD or death were assessed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 20 | 35
Months | 35.15 [33.05 to 37.13] | 21.75 [14.75 to 26.41]

6. Secondary Outcome: Investigator-assessed of Kaplan-meier Estimates of Progression-free Survival (PFS)
Description: PFS is defined as the interval of time between the date of the first administration of study treatment and the earlier of the date of disease progression (PD) and the date of death due to any cause. PD requires at least one of the following:new lesion or increase by >=50% from BL in LC, Ly, size of liver and spleen, PL >= 50% decrease from BL, or to <100,000/uL secondary to CLL, Hb decrease of >2 g/dL from BL or to <10 g/dL secondary to CLL, CLL- transformation. Response was determined according to the IWCLL updated NCI-WG guidelines 2008. Participants who have neither progressed or died at the time of analysis were censored at the date of the last adequate assessment. If there was more than 1 scheduled visit missed, PFS is censored at the last adequate assessment of response. An adequate assessment is defined as an assessment where the investigator determined a response of CR, CRi, nPR, PR, or stable disease (SD).
Time Frame: From the start of study treatment until earliest date of disease progression or death (up to 3 years after the last dose of study treatment)
Population: All Treated Subjects' (ATS) population. N= Progression or Death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 20 | 39
Months | 36.07 [34.00 to 38.05] | 22.54 [14.00 to 27.33]

7. Secondary Outcome: Investigator-assessed Kaplan-meier Estimates of Overall Survival
Description: OS is defined as the interval of time between the date of the first administration of study treatment and the date of death due to any cause. For participants who did not die, time of death was censored at the date of last contact.
Time Frame: From the start of study treatment to the date of death due to any cause (up to 3 years after the last dose of study treatment)
Population: All treated subjects. N= Death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 3 | 23
Months | NA [NA to NA] — Median was not available because over 50% of the all treated subjects were alive. | NA [NA to NA] — Median was not available because over 50% of the all treated subjects were alive.

8. Secondary Outcome: Investigator-Assessed Kaplan-Meier Estimates of Time to Progression
Description: Time to progression is defined as the time from the date of the first administration of study treatment to disease progression (PD). PD requires at least one of the following: new lesion or increase by >=50% from Baseline in lymphocytes (LC) with at least 5000 B-lymphocytes per microliter (5.0 x 10^9/L), lymphadenopathy (Ly), size of liver and spleen, platelets (PL) >= 50% decrease from Baseline, or to <100,000/uL secondary to CLL, hemoglobin (Hb) decrease of >2 g/dL from Baseline or to <10 g/dL secondary to CLL, CLL- transformation, cytopenia after treatment. Response was determined according to the IWCLL updated NCI-WG guidelines 2008.
Time Frame: From the start of study treatment to disease progression (up to 3 years after the last dose of study treatment)
Population: All treated subjects (ATS). This analysis includes patients who had progression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 19 | 35
Months | 36.0 [34.00 to 38.05] | 22.67 [16.07 to 28.58]

9. Secondary Outcome: Time to Next Therapy
Description: Time to next therapy is defined as the time from the date of the first administration of study treatment until the start of the next anti-CLL therapy.
Time Frame: From the start of study treatment until the start of the next anti-CLL therapy (up to 3 years after the last dose of study treatment)
Population: ATS Population. Only participants that took anti-CLL therapy were evaluated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 14 | 29
Months | 31.18 [17.25 to 37.03] | 16.82 [11.60 to 25.36]

10. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From first dose of study medication to 60 days after the last dose of study medication (if the event is considered as an AE), or up to 3 years after the last dose of study treatment or until the time of the next anti-CLL therapy, if considered a SAE
Population: Safety Population: all participants who received at least one dose of any study treatment (ofatumumab or bendamustine).
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  Any AE | 43 | 50
  Any SAE | 20 | 25

11. Secondary Outcome: Change From Baseline in the Immunoglobulin (Ig) Antibodies to End of Study Treatment
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. IgA, IgG, and IgM were measured in the blood samples of the participants. Baseline IgA, IgG, and IgM values are the last pre-dose assessment values performed on cycle 1 Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and end of study treatment (up to 30 months)
Population: Safety Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 38 | 43
Gram per liter
  IgA | 0.0768 (0.91109) | 0.0540 (0.23643)
  IgG | -0.714 (3.0614) | -1.246 (5.3194)
  IgM | -0.0490 (0.29267) | -0.0463 (0.16294)

12. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) CD5+CD19+ Cell Counts up to 36 Months
Description: CD5+ CD19+ cells were counted by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus. Baseline CD5+ CD19+ cell count value is the last pre-dose assessment values performed on cycle 1 Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline, 3-Month Follow-up to 36-Month Follow-up (in 3 months interval)
Population: ATS Population. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Cell per microliter
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Cell per microliter
  3 month F/U - Baseline (n=32, 31) | -72622.5 (104175.69) [9882 to 600336] | -40644.2 (36183.14) [2086 to 222187]
  6 month F/U - Baseline (n=30,28) | -61258.2 (42645.75) [0 to 899] | -45630.4 (40130.68) [0 to 4452]
  9 month F/U - Baseline (n=37,23) | -76688.7 (99375.55) [0 to 4055] | -49527.3 (40728.82) [0 to 17282]
  12 month F/U - Baseline (n=32,23) | -77884.8 (106795.41) | -43994.3 (39165.64)
  15 month F/U - Baseline (n=29,21) | -80997.6 (108950.32) | -39985.6 (36456.16)
  18 month F/U - Baseline (n=23,11) | -85837.7 (120525.82) | -31229.5 (28486.65)
  21 month F/U - Baseline (n=17,8) | -82180.6 (138188.36) | -52665.1 (42250.59)
  24 month F/U - Baseline (n=15,7) | -92850.6 (144547.27) | -37969.3 (26444.26)
  27 month F/U - Baseline (n=19, 6) | -82553.4 (129930.36) | -24824.8 (23700.40)
  30 month F/U - Baseline (n=15, 6) | -96903.7 (142080.38) | -30938.0 (28108.70)
  33 month F/U - Baseline (n=10, 3) | -65321.8 (40537.06) | -38216.3 (24864.31)
  36 month F/U - Baseline (n=8, 4) | -52087.1 (35735.07) | -30961.0 (25003.73)

13. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) CD5-CD19+ Cell Counts up to 36 Months
Description: CD5-CD19+ cells were counted by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus. Baseline CD5- CD19+ cell count value is the last pre-dose assessment values performed on cycle 1 Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline, 3-Month Follow-up to 36-Month Follow-up (in 3 months interval)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Cell per microliter
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Cell per microliter
  3 month F/U - Baseline (n= 32, 31) | -5800.8 (12693.09) [15 to 61395] | -2052.4 (5243.64) [7 to 85179]
  6 month F/U - Baseline (n= 30, 28) | -3921.1 (6959.20) [1 to 16] | -3822.8 (8449.80) [0 to 625]
  9 month F/U - Baseline (n= 37, 23) | -5969.7 (12277.21) [1 to 22] | -2288.4 (5724.47) [1 to 159]
  12 month F/U - Baseline (n= 32, 23) | -6756.8 (13009.04) | -4656.3 (9087.98)
  15 month F/U - Baseline (n= 29, 21) | -5323.6 (8727.91) | -4256.2 (9145.23)
  18 month F/U - Baseline (n= 23, 11) | -4677.9 (7677.12) | -5043.6 (10927.98)
  21 month F/U - Baseline (n= 17, 8) | -5224.2 (8477.84) | -275.1 (449.28)
  24 month F/U - Baseline (n= 15, 7) | -4522.7 (7562.59) | -224.0 (447.47)
  27 month F/U - Baseline (n= 19, 6) | -7259.0 (10162.96) | -3870.5 (8960.80)
  30 month F/U - Baseline (n= 15, 6) | -7673.6 (10238.82) | -3964.3 (8918.40)
  33 month F/U - Baseline (n= 10, 3) | -9511.2 (11834.25) | -206.0 (215.84)
  36 month F/U - Baseline (n= 8, 4) | -8430.1 (13019.82) | -5693.0 (10969.00)

14. Secondary Outcome: Number of Participants Who Were Negative or Positive for Minimal Residual Disease (MRD) and Achieved a Bone Marrow Biopsy Confirmed Complete Response (CR) up to 36-Month Follow-up
Description: MRD refers to small number of leukemic cells that remain in the participant during treatment or after treatment at the time the participant achieved a confirmed CR. MRD analysis was performed for the partcipants who were suspected of achieving a primary endpoint CR. Analysis of CD5+ CD19+ was performed on the bone marrow aspirate sample obtained no sooner than 2 months following the last dose of study treatment. MRD results were reported as negative or positive. The absence of MRD (negative MRD) is defined as less than one CLL cell per 10000 leukocytes.
Time Frame: 3 month follow up to the 36 Month Follow-up (in 3 month interval)
Population: ATS Population. Number of subjects who had CR with bone marrow confirmation are included. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 16 | 4
Participants
  3 month F/U, MRD Positive (n=16 , 4) | 7 | 4
  3 month F/U, MRD Negative (n=16 , 4) | 9 | 0
  6 month F/U, MRD Positive (n=8 , 2) | 1 | 1
  6 month F/U, MRD Negative (n=8 , 2) | 7 | 1
  9 month F/U, MRD Positive (n=11 , 2) | 3 | 1
  9 month F/U, MRD Negative (n=11 , 2) | 8 | 1
  12 month F/U, MRD Positive (n=9 , 2) | 1 | 1
  12 month F/U, MRD Negative (n=9 , 2) | 8 | 1
  15 month F/U, MRD Positive (n=9 , 2) | 3 | 1
  15 month F/U, MRD Negative (n=9 , 2) | 6 | 1
  18 month F/U, MRD Positive (n=6 , 1) | 1 | 0
  18 month F/U, MRD Negative (n=6 , 1) | 5 | 1
  21 month F/U, MRD Positive (n=7, 1) | 2 | 0
  21 month F/U, MRD Negative (n=7 , 1) | 5 | 1
  24 month F/U, MRD Positive (n=6 , 1) | 0 | 0
  24 month F/U, MRD Negative (n=6 , 1) | 6 | 1
  27 month F/U, MRD Positive (n=3 , 1) | 0 | 0
  27 month F/U, MRD Negative (n=3 , 1) | 3 | 1
  30 month F/U, MRD Positive (n=4 , 1) | 1 | 0
  30 month F/U, MRD Negative (n=4 , 1) | 3 | 1
  33 month F/U, MRD Positive (n=4 , 1) | 1 | 0
  33 month F/U, MRD Negative (n=4 , 1) | 3 | 1
  36 month F/U, MRD Positive (n=2 , 1) | 0 | 0
  36 month F/U, MRD Negative (n=2 , 1) | 2 | 1

15. Secondary Outcome: Number of Participants Who Received no Transfusion or at Least One Transfusion During the Study
Description: Participants who received no transfusion and at least one transfusion during the study are presented. Participants who took any blood products are counted in this table.
Time Frame: From start of treatment until earliest date of disease progression or death (up to 3 years after the last dose of study treatment)
Population: Safety Population: All subjects who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  No transfusions | 38 | 33
  At least one transfusion | 6 | 20

16. Secondary Outcome: Number of Participants With Autoimmune Hemolytic Anaemia (AIHA) Disease
Description: AIHA is a disease where the body's immune system fails to recognize red blood cells as "self" and begins destroying these red blood cells. The number of participants diagnosed with AIHA are presented.
Time Frame: as for outcome 10
Population: Safety Population All subjects who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants | 0 | 1

17. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Myelosuppression (Anemia, Neutropenia, and Thrombocytopenia), as Assessed by the Investigator
Description: Participants with a Grade 3 or Grade 4 myelosuppression (anemia, neutropenia, and thrombocytopenia) are presented. Myelosuppression is defined as the decrease in the ability of the bone marrow to produce blood cells. AEs were graded according to NCI common terminology criteria for adverse events (CTCAE) grade, version 4.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: From the first dose of study medication to 60 days after the last dose of study medication
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  Neutropenia/Febrile neutropenia, Grade 3 | 8 | 27
  Neutropenia/Febrile Neutropenia, Grade 4 | 9 | 16
  Thrombocytopenia, Grade 3 | 1 | 2
  Thrombocytopenia, Grade 4 | 0 | 2
  Anemia, Grade 3 | 1 | 0
  Anemia, Grade 4 | 0 | 0

18. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Adverse Event of Infection
Description: Participants with the indicated Grade 3 or Grade 4 adverse event of infection are presented. AEs were graded according to the NCI CTCAE grade, version 4.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: as for outcome 10
Population: Safety Population: All subjects who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants | 5 | 10

19. Secondary Outcome: Number of Participants With the Indicated Constitutional or B-symptoms
Description: Participants with the indicated constitutional or B-symptoms (night sweats, weight loss, fever or extreme fatigue) were presented for different time points.
Time Frame: Screening (SCR), Cycle 3 Day 1 (C3D1), Cycle 6 Day 1 (C6D1), 12, 24 and 36 Month Follow-up (F/U)
Population: Safety Population: All subjects who receive at least one dose of study medication. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  SCR, night sweats, n =44, 52 | 19 | 22
  SCR, weight loss, n=44, 52 | 4 | 5
  SCR, fever, n=44, 52 | 1 | 2
  SCR, extreme fatigue, n=44, 52 | 14 | 15
  C3D1, night sweats, n =42, 49 | 5 | 2
  C3D1, weight loss, n=42, 49 | 0 | 2
  C3D1, fever, n=42, 49 | 0 | 0
  C3D1, extreme fatigue, n=42, 49 | 2 | 4
  C6D1, night sweats, n =39, 47 | 0 | 1
  C6D1, weight loss, n =39, 47 | 0 | 0
  C6D1, fever, n =39, 47 | 0 | 0
  C6D1, extreme fatigue, n =39, 47 | 0 | 1
  12 Month F/U, night sweats, n =39, 29 | 0 | 0
  12 Month F/U, weight loss, n =39, 29 | 1 | 0
  12 Month F/U, fever, n =39, 29 | 0 | 0
  12 Month F/U, extreme fatigue, n =39, 29 | 0 | 0
  24 Month F/U, night sweats, n =29, 17 | 0 | 0
  24 Month F/U, weight loss, n=29, 17 | 0 | 0
  24 Month F/U, fever, n=29, 17 | 0 | 0
  24 Month F/U, extreme fatigue, n=29, 17 | 1 | 0
  36 Month F/U, night sweats, n =21, 9 | 0 | 0
  36 Month F/U, weight loss, n=21, 9 | 0 | 0
  36 Month F/U, fever, n=21, 9 | 0 | 0
  36 Month F/U, extreme fatigue, n=21, 9 | 0 | 0

20. Secondary Outcome: Number of Participants With the Indicated Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: The ECOG performance status scales and criteria are used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. Grade 0, fully active, able to carry on all pre-disease performance without restriction. Grade 1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. Grade 2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about more than 50% of waking hours. Grade 3, capable of only limited selfcare; confined to bed or chair more than 50% of waking hours. Grade 4, completely disabled; cannot carry on any selfcare; totally confined to bed or chair. Grade 5, dead.
Time Frame: Baseline (BL), Cycle 3 Day 1 (C3D1), Cycle 6 Day 1 (C6D1), 12, 24 and 36 month follow up (F/U)
Population: Safety Population. All subjects who receive at least one dose of study medication.. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  BL, Score of 0, n=44, 53 | 16 | 23
  BL, Score of 1, n=44, 53 | 28 | 29
  BL, Score of 2, n=44, 53 | 0 | 1
  BL, Score of 3, n=44, 53 | 0 | 0
  BL, Score of 4-5, n=44, 53 | 0 | 0
  C3D1, Score of 0, n=42, 48 | 17 | 27
  C3D1, Score of 1, n=42, 48 | 25 | 21
  C3D1, Score of 2, n=42, 48 | 0 | 0
  C3D1, Score of 3, n=42, 48 | 0 | 0
  C3D1, Score of 4-5, n=42, 48 | 0 | 0
  C6D1, Score of 0, n=38, 47 | 19 | 27
  C6D1, Score of 1, n=38, 47 | 19 | 19
  C6D1, Score of 2, n=38, 47 | 0 | 1
  C6D1, Score of 3, n=38, 47 | 0 | 0
  C6D1, Score of 4-5, n=38, 47 | 0 | 0
  12 Month F/U, Score of 0, n=39, 28 | 24 | 19
  12 Month F/U, Score of 1, n=39, 28 | 14 | 8
  12 Month F/U, Score of 2, n=39, 28 | 1 | 1
  12 Month F/U, Score of 3, n=39, 28 | 0 | 0
  12 Month F/U, Score of 4-5, n=39, 28 | 0 | 0
  24 Month F/U, Score of 0, n=28, 16 | 16 | 13
  24 Month F/U, Score of 1, n=28, 16 | 11 | 3
  24 Month F/U, Score of 2, n=28, 16 | 1 | 0
  24 Month F/U, Score of 3, n=28, 16 | 0 | 0
  24 Month F/U, Score of 4-5, n=28, 16 | 0 | 0
  36 Month F/U, Score of 0, n=21, 9 | 15 | 8
  36 Month F/U, Score of 1, n=21, 9 | 5 | 1
  36 Month F/U, Score of 2, n=21, 9 | 1 | 0
  36 Month F/U, Score of 3, n=21, 9 | 0 | 0
  36 Month F/U, Score of 4-5, n=21, 9 | 0 | 0

21. Secondary Outcome: Number of Participants With Confirmed Positive Response for Human Anti-human Antibodies (HAHA) at the Indicated Time Points
Description: The presence of HAHA in human serum was determined using a validated electrochemiluminescent assay in a multi-tier assay format. All samples were first assessed in a screening (SCR) assay, and the potential positive (Pos) samples were further tested in the confirmation (CNF) assays. Confirmed positives were reported as HAHA positive and titer was determined for each positive sample. The drug tolerance of the HAHA assay is 200 microgram/milliliter (µg/mL); thus, samples that tested negative in the assay and had ofatumumab concentrations no more than 200 µg/mL were considered as conclusive negative (C Neg) results.
Time Frame: Cycle 1 Day 1 (C1D1), Cycle 6 Day 1 (C6D1), 6-Month Follow-up (F/U), and any post-dose time point
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  C1D1, n=41, 53 | 0 | 0
  C6D1, n=34, 43 | 0 | 0
  6-Month F/U, n=35, 37 | 0 | 0
  Any post dose time, n=42, 47 | 0 | 0

22. Secondary Outcome: Maximum Decrease in Sum of the Product of the Diameter (SPD) From Baseline in Participants With Lymphadenopathy at Baseline
Description: Lymph nodes were evaluated by physical examination which involved recording the diameter in two planes (sum of the product of the diameter [SPD]) of the largest palpable node in each of the following sites: cervical, axillary, supraclavicular, inguinal and femoral. Lymphadenopathy is defined as lymph nodes with the largest diameter greater than 1.5 centimeters. The maximum reduction in SPD from Baseline at C2D1, C3D1, C4D1, C5D1, C6D1, 3-Month F/U, 6-Month F/U and 9-Month F/U are provided.
Time Frame: Baseline, Cycle 2 Day 1 (C2D1), Cycle 3 Day 1 (C3D1), Cycle 4 Day 1 (C4D1), Cycle 5 Day 1 (C5D1), Cycle 6 Day 1 (C6D1), 3-Month Follow-Up (F/U), 6-Month F/U and 9-Month F/U
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: cm^2 (centimeters squared)
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
cm^2 (centimeters squared)
  C2D1, n=34, 35 | -83.5 (23.69) | -77.3 (31.62)
  C3D1, n=32, 35 | -92.1 (20.17) | -90.9 (17.18)
  C4D1, n=32, 35 | -99.1 (2.67) | -94.6 (11.56)
  C5D1, n=29, 35 | -99.6 (1.22) | -96.2 (8.95)
  C6D1, n=30, 33 | -99.6 (2.28) | -97.0 (7.78)
  3-Month F/U, n=33, 32 | -99.2 (3.64) | -95.9 (19.17)
  6-Month F/U, n=3, 1 | -100.0 (0.00) | -100.0 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the standard deviation cannot be calculated.
  9-Month F/U, n=1, 0 | -68.4 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

23. Secondary Outcome: Number of Participants With the Indicated Reduction in Organomegaly (Spleen and Liver)
Description: Organomegaly is the abnormal enlargement of organs. Physical examination of the liver (L) and spleen (S) were done at Screening (SCR), C3D1, C6D1, 12-Month F/U, 24-Month F/U and 36-Month F/U. The result of the physical examination of the liver (L) and spleen (S) was presented as normal (NOR), enlarged (EL) and not assessed (NOA).
Time Frame: Screening (Scr), Cycle 3 Day 1 (C3D1), Cycle 6 Day 1 (C6D1), 12, 24 and 36 -Month Follow-Up (F/U)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  SCR, S, NOR, n=44, 50 | 23 | 31
  SCR, S, EL, n=44, 50 | 21 | 19
  SCR, S, NOA, n=44, 50 | 0 | 0
  SCR, L, NOR, n=44, 51 | 38 | 41
  SCR, L, EL, n=44, 51 | 6 | 9
  SCR, L, NOA, n=44, 51 | 0 | 1
  C3D1, S, NOR, n=42, 48 | 37 | 41
  C3D1, S, EL, n=42, 48 | 5 | 6
  C3D1, S, NOA, n=42, 48 | 0 | 1
  C3D1, L, NOR, n=42, 48 | 38 | 42
  C3D1, L, EL, n=42, 48 | 4 | 5
  C3D1, L, NOA, n=42, 48 | 0 | 1
  C6D1, S, NOR, n=39, 46 | 39 | 43
  C6D1, S, EL, n=39, 46 | 0 | 2
  C6D1, S, NOA, n=39, 46 | 0 | 1
  C6D1, L, NOR, n=39, 46 | 37 | 44
  C6D1, L, EL, n=39, 46 | 2 | 0
  C6D1, L, NOA, n=39, 46 | 0 | 2
  12 Month F/U, S, NOR, n=39, 29 | 39 | 28
  12 Month F/U, S, EL, n=39, 29 | 0 | 1
  12 Month F/U, S, NOA, n=39, 29 | 0 | 0
  12 Month F/U, L, NOR, n=39, 29 | 38 | 28
  12 Month F/U, L, EL, n=39, 29 | 1 | 1
  12 Month F/U, L, NOA, n=39, 29 | 0 | 0
  24 Month F/U, S, NOR, n=29, 17 | 29 | 16
  24 Month F/U, S, EL, n=29, 17 | 0 | 1
  24 Month F/U, S, NOA, n=29, 17 | 0 | 0
  24 Month F/U, L, NOR, n=29, 17 | 29 | 16
  24 Month F/U, L, EL, n=29, 17 | 0 | 1
  24 Month F/U, L, NOA, n=29, 17 | 0 | 0
  36 Month F/U, S, NOR, n=21, 9 | 21 | 9
  36 Month F/U, S, EL, n=21, 9 | 0 | 0
  36 Month F/U, S, NOA, n=21, 9 | 0 | 0
  36 Month F/U, L, NOR, n=21, 9 | 21 | 9
  36 Month F/U, L, EL, n=21, 9 | 0 | 0
  36 Month F/U, L, NOA, n=21, 9 | 0 | 0

24. Secondary Outcome: Number of Participants With the Indicated Cytogenetics Testing at Baseline Who Also Had a Clinical Response After Last Dose of Study Treatment
Description: Cytogenetics refers to the study of numerical and structural chromosomal abnormalities. Cytogenetics (analyzed by fluorescent in situ hybridization [FISH]) of 17p deletion, 11q deletion, 17p or 11q deletions, 6q- or +12q or 13q- deletions, and no aberration at Baseline were summarized by clinical responses after the last dose of study treatment. Clinical responses included complete remission (CR), nodular partial remission (nPR), complete response with incomplete bone marrow Recovery (CRi), partial remission (PR), disease progression (PD), and stable disease (SD). The participants with a PR, CRi, PR or nPR are called responders and the participants with SD and PD are called non-responders.
Time Frame: From the start of study treatment until earliest date of disease progression or death (up to up to 3 months following last dose of study treatment)
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  17p-, CR, n=2, 6 | 0 | 0
  17p-, CRi, n=2, 6 | 0 | 0
  17p-, nPR, n=2, 6 | 0 | 0
  17p-, PR, n=2, 6 | 0 | 1
  17p-, SD, n=2, 6 | 1 | 3
  17p-, PD, n=2, 6 | 0 | 2
  11q-, CR, n=8, 15 | 3 | 1
  11q-, CRi, No, n=8, 15 | 0 | 0
  11q-, nPR, n=8, 15 | 1 | 3
  11q-, PR, n=8, 15 | 4 | 7
  11q-, SD, n=8, 15 | 0 | 1
  11q-, PD, n=8, 15 | 0 | 3
  17p- or 11q-, CR, n=10, 20 | 3 | 1
  17p- or 11q-, CRi, n=10, 20 | 0 | 0
  17p- or 11q-, nPR, n=10, 20 | 1 | 3
  17p- or 11q-, PR, n=10, 20 | 4 | 8
  17p- or 11q-, SD, n=10, 20 | 1 | 3
  17p- or 11q-, PD, n=10, 20 | 0 | 5
  6q- or +12q or 13q-, CR, n=20, 24 | 11 | 3
  6q- or +12q or 13q-, CRi, n=20, 24 | 1 | 2
  6q- or +12q or 13q-, nPR, n=20, 24 | 1 | 4
  6q- or +12q or 13q-, PR, n=20, 24 | 7 | 10
  6q- or +12q or 13q-, SD, n=20, 24 | 0 | 2
  6q- or +12q or 13q-, PD, n=20, 24 | 0 | 2
  No aberration, CR, n= 14, 8 | 5 | 2
  No aberration, CRi, n= 14, 8 | 2 | 0
  No aberration, nPR, n= 14, 8 | 3 | 1
  No aberration, PR, n= 14, 8 | 4 | 4
  No aberration, SD, n= 14, 8 | 0 | 0
  No aberration, PD, n= 14, 8 | 0 | 1

25. Secondary Outcome: Number of Participants With the Indicated Beta 2 Microglobulin (B2M) at Baseline Who Also Had a Clinical Response After the Last Dose of Study Treatment
Description: Participants with B2M concentration of <=4000 µg/L and >4000 µg/L at Baseline and who had clinical response after the last dose of study treatment were provided. Clinical responses included complete remission (CR), complete response with incomplete bone marrow Recovery (CRi), nodular partial remission (nPR), and partial remission (PR), disease progression (PD), and stable disease (SD). The participants with a PR, CRi, PR or nPR are called responders and the participants with SD and PD are called non-responders.
Time Frame: as for outcome 24
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  <= 4000 µg/L, CR, n=23, 24 | 9 | 3
  <= 4000 µg/L, CRi, n=23, 24 | 3 | 2
  <= 4000 µg/L, nPR, n=23, 24 | 4 | 6
  <= 4000 µg/L, PR, n=23, 24 | 7 | 9
  <= 4000 µg/L, SD, n=23, 24 | 0 | 2
  <= 4000 µg/L, PD, n=23, 24 | 0 | 2
  > 4000 µg/L, CR, n=17, 29 | 9 | 3
  > 4000 µg/L, CRi, n=17, 29 | 0 | 0
  > 4000 µg/L, nPR, n=17, 29 | 1 | 2
  > 4000 µg/L, PR, n=17, 29 | 6 | 14
  > 4000 µg/L, SD, n=17, 29 | 0 | 3
  > 4000 µg/L, PD, n=17, 29 | 0 | 6

26. Secondary Outcome: Number of Participants With the Indicated Immunoglobulin Heavy Chain Variable Region (IgVH) Testing at Baseline Who Also Had a Clinical Response After Last Dose of Study Treatment
Description: Participants with IgVH mutation results as mutated and unmutated status and clinical response after last dose of study treatment were provided. Clinical responses included complete remission (CR), complete response with incomplete bone marrow recovery (CRi), nodular partial remission (nPR), partial remission (PR), disease progression (PD), and stable disease (SD). The participants with a PR, CRi, PR or nPR are called responders and the participants with SD and PD are called non-responders.
Time Frame: as for outcome 24
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  IgVH Mutated (<=98 %), CR, n=12, 13 | 6 | 4
  IgVH Mutated (<=98 %), CRi, n=12, 13 | 2 | 0
  IgVH Mutated (<=98 %), nPR, n=12, 13 | 0 | 4
  IgVH Mutated (<=98 %), PR, n=12, 13 | 4 | 2
  IgVH Mutated (<=98 %), SD, n=12, 13 | 0 | 0
  IgVH Mutated (<=98 %), PD, n=12, 13 | 0 | 3
  IgVH unmutated (>98%), CR, n=23, 34 | 11 | 1
  IgVH unmutated (>98%), CRi, n=23, 34 | 1 | 2
  IgVH unmutated (>98%), nPR, n=23, 34 | 5 | 4
  IgVH unmutated (>98%), PR, n=23, 34 | 5 | 18
  IgVH unmutated (>98%), SD, n=23, 34 | 0 | 5
  IgVH unmutated (>98%), PD, n=23, 34 | 0 | 3

27. Secondary Outcome: Number of Participants With Zeta-chain-associated Protein Kinase (ZAP) 70 Testing at Baseline Who Also Had a Clinical Response After Last Dose of Study Treatment
Description: ZAP-70 is a protein normally expressed near the surface membrane of T cells and natural killer cells. ZAP-70 in B cells is used as a prognostic marker in identifying different forms of CLL. Participants with ZAP-70 testing results intermediate (Int), positive (Pos) and negative (Neg) at Baseline and who had a clinical response after last dose of study treatment are provided. Clinical responses included complete remission (CR), complete response with incomplete bone marrow recovery (CRi), nodular partial remission (nPR), partial remission (PR), disease progression (PD), and stable disease (SD). The participants with a PR, CRi, PR or nPR are called responders and the participants with SD and PD are called non-responders.
Time Frame: From the start of study treatment until earliest date of disease progression or death (up to 3 months following last dose of study treatment)
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 36 | 44
Participants
  ZAP-70, Int, CR, n=6, 6 | 1 | 1
  ZAP-70, Int, CRi, n=6, 6 | 0 | 0
  ZAP-70, Int, nPR, n=6, 6 | 0 | 0
  ZAP-70, Int, PR, n=6, 6 | 3 | 3
  ZAP-70, Int, PD, n=6, 6 | 0 | 1
  ZAP-70, Int, SD, n=6, 6 | 1 | 0
  ZAP-70, Neg, CR, n=2, 2 | 1 | 0
  ZAP-70, Neg, CRi, n=2, 2 | 0 | 0
  ZAP-70, Neg, nPR, n=2, 2 | 0 | 0
  ZAP-70, Neg, PR, n=2, 2 | 1 | 2
  ZAP-70, Neg, PD, n=2, 2 | 0 | 0
  ZAP-70, Neg, SD, n=2, 2 | 0 | 0
  ZAP-70, Pos, CR, n=36, 44 | 17 | 5
  ZAP-70, Pos, CRi, n=36, 44 | 3 | 2
  ZAP-70, Pos, nPR, n=36, 44 | 5 | 8
  ZAP-70, Pos, PR, n=36, 44 | 11 | 17
  ZAP-70, Pos, PD, n=36, 44 | 0 | 7
  ZAP-70, Pos, SD, n=36, 44 | 0 | 5

28. Secondary Outcome: Number of Participants With an Adverse Event of Any Infusion Reactions (IR) or Serious Infusion Reactions (SIR)
Description: An Infusion reaction is defined as events occurring after the beginning of an infusion of ofatumumab or within 24 hours following the end of an infusion of bendamustine.
Time Frame: From the first dose of study medication to 60 days after the last dose of study medication (up to 24 hours after last dose of study treatment)
Population: Safety Population: All subjects who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Bendamustine 90 mg/m^2 | Ofatumumab + Bendamustine 70 mg/m^2
Number analyzed (Participants) | 44 | 53
Participants
  Any ofatumumab only IR | 30 | 34
  Any ofatumumab only SIR | 3 | 4
  Any ofatumumab plus bendamustine IR | 30 | 35
  Any ofatumumab plus bendamustine SIR | 4 | 4

ADVERSE EVENTS:
Time Frame: From the first dose of study medication to 60 days after the last dose of study medication (if the event is considered as an AE), or up to 3 years after the last dose of study treatment or until the time of the next anti-CLL therapy, if considered a SAE.
Description: Serious adverse events (SAEs) and and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of any study drug (ofatumumab or bendamustine).
Groups:
- Ofatumumab + Bendamustine 70mg/m^2: Participants with relapsed CLL received IV infusions of ofatumumab in combination with bendamustine IV infusions for 6 cycles; each cycle comprised of 28 days. Participants received ofatumumab administered at 300 mg on Day 1, 1000 mg on Day 8 of cycle 1 and 1000 mg on Day 1 of cycles 2, 3, 4, 5 and 6. Bendamustine was administered at 70 mg/m^2 on Days 1 and 2 of each cycle (6 cycles).
- Ofatumumab + Bendamustine 90mg/m^2: Participants with previously untreated CLL received IV infusions of ofatumumab in combination with bendamustine IV infusions for 6 cycles; each cycle comprised of 28 days. Participants received ofatumumab administered at 300 mg on Day 1, 1000 mg on Day 8 of cycle 1 and 1000 mg on Day 1 of cycles 2, 3, 4, 5 and 6. Bendamustine was administered at 90 mg/m^2 on Days 1 and 2 of each cycle (6 cycles).
Arm/Group | Ofatumumab + Bendamustine 70mg/m^2 | Ofatumumab + Bendamustine 90mg/m^2
Serious Adverse Events (participants affected / at risk) | 25/53 | 20/44
Other Adverse Events (participants affected / at risk) | 49/53 | 40/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Bendamustine 70mg/m^2 (N=53) | Ofatumumab + Bendamustine 90mg/m^2 (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Anaphylactic reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Erysipelothrix infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Bendamustine 70mg/m^2 (N=53) | Ofatumumab + Bendamustine 90mg/m^2 (N=44)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 32 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 7
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 16 | 19
Vomiting (Gastrointestinal disorders) | 4 | 5
Asthenia (General disorders) | 3 | 5
Chills (General disorders) | 3 | 5
Fatigue (General disorders) | 8 | 7
Malaise (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 4 | 3
Pyrexia (General disorders) | 8 | 10
Bronchitis (Infections and infestations) | 3 | 2
Herpes simplex (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Urinary tract infection (Infections and infestations) | 2 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 3
Blood creatinine increased (Investigations) | 3 | 3
Weight decreased (Investigations) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 6 | 6
Insomnia (Psychiatric disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 5 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 7 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 6
Flushing (Vascular disorders) | 5 | 1
Phlebitis (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.